CLINICAL TRIAL: NCT05175014
Title: Determining Whether Mass Campaigns With Fractional Dose PCV10 Would Accelerate Herd Protection Against Pneumococcal Transmission in Sub-Saharan Africa
Brief Title: Mass Campaigns With Fractional Dose Pneumococcal Vaccines in Sub-Saharan Africa (fPCV)
Acronym: fPCV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Epicentre (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other); Kenya Medical Research Institute (Other); Universite Abdou Moumouni de Niamey, Niger (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: fPCV
Record Dates: First submitted 2021-12-13; First posted 2022-01-03 (Actual); Results first posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-11

CONDITIONS: Pneumococcal Carriage

STUDY DESIGN:
Intervention Model Description: A Phase IV, 3-arm, observer-blinded, cluster-randomized controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Vaccinators will not be blinded, but participants will not know vaccine dosage allocation. Laboratory staff (outcome assessors) will be blinded to their group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Single full dose of PCV 10 (Experimental): 27 clusters randomized to receive a vaccination campaign with the full dose.
  Interventions: Biological: PCV10 full dose
- Single fractional dose of PCV10 (1/5) (Experimental): 27 clusters randomized to receive a vaccination campaign with the fractional dose (1/5).
  Interventions: Biological: PCV10 fractional dose
- Control Group (No Intervention): 9 clusters randomized to the control arm.

INTERVENTIONS:
Biological: PCV10 full dose — Mass vaccination campaign with one single dose PCV10 vaccine administered as a full dose.
  Arms: Single full dose of PCV 10
Biological: PCV10 fractional dose — Mass vaccination campaign with one single dose PCV10 vaccine administered as a fractional dose.
  Arms: Single fractional dose of PCV10 (1/5)

SUMMARY:
The aim of this study is to assess the impact of a mass campaign with a single, fractional dose of Pneumosil®, a PCV10, on VT carriage. A 20% fractional dose (1/5th) will be used as a practical formulation to prepare and administer. This study will assess whether the impact of a single fractional dose mass campaign on carriage is non-inferior to a single full dose mass campaign in a cluster randomized trial in a low coverage setting in Niger. The results would provide evidence of the population-level direct and indirect impact of fractional dose in older children which will be completed by mathematical modelling, to inform the policy debate regarding PCV dosing schedules in different contexts. This trial and the modelling exercises that follow, would allow for larger scale evaluation of fractional dose PCV strategies in multiple contexts.

DETAILED DESCRIPTION:
In 2015, there were an estimated 8.9 million cases (uncertainty range 7.7-10.6 million) of clinical pneumococcal pneumonia globally, with 2.4 million cases estimated in Africa alone (uncertainty range 2.1-3.1 million). These figures represent a global reduction of 37% from 14.2 million cases (12.3 million-16.9 million) in 2000. However, pneumococcal disease continues to be a leading cause of severe disease and death representing 10% of all death in children under 5 years of age (1). These deaths occur disproportionally in low- and middle-income countries (LMICs), with approximately 50% of global pneumococcal deaths estimated to occur in 4 countries: India, Nigeria, Pakistan and the Democratic Republic of Congo.

Vaccination campaigns targeting children up to 5 years of age have an effect in the reduction of VT carriage disease. However, in crises or settings with high prevalence of malnutrition, the high pneumococcal carriage prevalence is likely to extend to older age groups. Single dose vaccination of a larger age group might be needed to control VT circulation. Currently, for GAVI-supported countries such as Niger, PCV13 vaccine has a cost of US$3 per dose. Pneumosil®, a PCV10 manufactured by Serum institute of India Ltd has the lowest price of all WHO prequalified vaccines, at US$2 per dose.

Mass campaigns targeting large groups require many doses and might not be sustainable over time. Fractional doses of PCV could be a solution to overcome the high PCV costs, increase vaccine access and expand vaccination benefits through alternative strategies. The study population (ages 1-9) stems from an LSHTM modelling study.

Objectives of the study Primary objective: evaluate whether the full dose of PCV is superior to the absence of vaccine and then if a single 20% dose of PCV is non-inferior to a full dose in carriage reduction.

Secondary objectives:

* To measure the age-stratified prevalence of NP carriage of S. pneumoniae in children 1-9 years of age in the study area.
* To determine the impact of a mass vaccination campaign with one full dose of PCV in children 1 to 9 years of age on VT pneumococci carriage 6 months after vaccination
* To assess the occurrence of adverse events (AE) and serious adverse events (SAE) during 28 days after administration of fractional and full doses and SAEs throughout the duration of follow-up
* To model the potential impact of fractional dose PCV campaigns in other contexts using the results of the clinical trial.
* To develop recommendations on how a potential future fractional dose PCV mass campaign could be successfully planned, communicated, delivered, and integrated into national immunization programmes using qualitative analysis.

Note: the 1-9 years age group targeted for the mass campaign is based on data from a model in Kilifi, Kenya. Baseline carriage survey data together with data will be used on interactions between age groups and PCV coverage data collected during the baseline survey, to estimate the age group that should be targeted for vaccination.

Methodology A cluster-randomized, blinded, non-inferiority trial will be implemented in rural villages of the Madarounfa District of Niger. Clusters will be randomized to full dose, fractional dose or control arm in 2:2:1 allocation ratio. Clusters will be composed of a village or group of neighbouring villages that share a school or market. Stratified randomization will be used to consider size of clusters and proximity to health centre. Vaccination will target all children aged approximately 1 to 9 years of age residing in the selected villages Prior to the mass vaccination campaign, a cross-sectional survey will be implemented to estimate community-level carriage of VT pneumococci, as well as to collect data on household composition, social interactions and PCV vaccination coverage.

ELIGIBILITY:
For participation in pneumococcal carriage surveys:

Inclusion criteria:

1. Aged 1-9 years
2. Residing in the villages included in the study
3. Parent or caretaker provides informed consent for the child to participate in the study

Exclusion criteria:

1. Head or facial injuries that contraindicate nasopharyngeal swabbing
2. Any condition or criteria, including acute or chronic clinically significant abnormality that in the opinion of the investigator might compromise the wellbeing of the participant or interfere with the outcome of the study

For participation in mass vaccination campaigns (with full or fractional dose PCV10)

Inclusion criteria:

1. Aged 1-9 years
2. Residing in the villages included in the study and allocated to vaccination
3. Head of the household or main caretaker provides consent for the child to be vaccinated

Exclusion criteria:

1. Hypersensitivity to any component of the vaccine, including diphtheria toxoid
2. Vaccination with a PCV vaccine within the previous 4 weeks, as there should be a minimum of 4 weeks between doses
3. Moderate or severe febrile illness (temperature ≥39°C) is a temporal contraindication and the child should not be vaccinated until improvement
4. Any condition or criteria, including acute or chronic clinically significant abnormality that in the opinion of the clinical staff might compromise the wellbeing of the volunteer

Ages: 1 Year to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 44618 (Actual)
Dates: Start 2021-12-30 (Actual); Primary Completion 2023-03-14 (Actual); Study Completion 2023-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Rebecca Grais, Study Director — Epicentre Research Department Director; Dr. Matthew Coldiron, Principal Investigator — Epicentre Research Department Investigator; Dr. Issaka Soumana, Principal Investigator — Epicentre Niger Research Center Assistant Manager
Locations (1):
- Epicentre, Maradi, Niger

IPD SHARING:
Plan to Share IPD: Yes
IPD will consist of sociodemographic data collected in baseline and post-vaccination surveys, as well as results of pneumococcal isolation and serotyping.
Time Frame: De-identified IPD will be available after final data collection and cleaning, and once laboratory quality control procedures have been conducted.
Access Criteria: Any interested party may request access to the data for the purposes of secondary analysis or meta-analysis. The process for requesting data, and the criteria upon which requests will be judged are described in Epicentre Standard Operating Procedures.

REFERENCES:
- [Derived] Coldiron ME, Soumana I, Baudin E, Langendorf C, Mamiafo Tchoula C, Brah S, Karani A, Gallagher KE, Kagucia EW, Scott JAG, Grais RF. Effect of mass campaigns with full and fractional doses of pneumococcal conjugate vaccine (Pneumosil) on the reduction of nasopharyngeal pneumococcal carriage in Niger: a three-arm, open-label, cluster-randomised trial. Lancet Infect Dis. 2025 Jun;25(6):634-642. doi: 10.1016/S1473-3099(24)00719-9. Epub 2025 Jan 8. PMID 39798587

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In the lead-in to the study, the total number of participants living in the 63 clusters was estimated to be approximately 32000. After study initiation, more accurate population figures were obtained, leading to the actual 44618 participants described in the reported results.
Units Other Than Participants: Clusters
Period: Overall Study
Arm/Group | Single Full Dose of PCV 10 | Single Fractional Dose of PCV10 (1/5) | Control Group
Started | 20091; 27 Clusters | 18821; 27 Clusters | 5706; 9 Clusters
Completed | 20091; 27 Clusters | 18821; 27 Clusters | 5706; 9 Clusters
Not Completed | 0; 0 Clusters | 0; 0 Clusters | 0; 0 Clusters

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Single Full Dose of PCV 10 | Single Fractional Dose of PCV10 (1/5) | Control Group | Total
Number analyzed (Participants) | 955 | 948 | 320 | 2223
Age, Continuous [Mean (Standard Deviation); unit: years] — Age of participants randomly selected from overall study population to participate in baseline nasopharyngeal carriage survey
  years | 4.5 (0.5) | 4.3 (0.6) | 4.5 (0.6) | 4.4 (0.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Sex breakdown of participants randomly selected from overall study population to participate in baseline nasopharyngeal carriage survey
  Participants
    Female | 482 | 473 | 157 | 1112
    Male | 473 | 475 | 163 | 1111
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Niger | 955 | 948 | 320 | 2223
Baseline prevalence of VT pneumococcal carriage [Number; unit: Percentage of participants] | 15.6 | 17.9 | 18.8 | 17.0

OUTCOME MEASURES:

1. Primary Outcome: Effect of a Single Dose PCV10 Campaign in the Reduction of VT Carriage
Description: The effect of a single dose PCV10 campaign in the reduction of VT carriage will be assessed by: first, assessing the superiority of a campaign using full doses of PCV10 compared to control group without vaccination; and second, by establishing the non-inferiority of a campaign using fractional doses of PCV10 compared to a campaign using full doses. NP carriage will be measured in the 3 study arms (full dose arm, fractional dose arm and control arm) in a baseline survey implemented prior to the vaccination campaign and in a post-vaccination survey. The NP carriage of VT S. pneumoniae will be measured as the proportion of participants that are colonized with any of the 10 serotypes covered by PCV10 at each time point. The reduction in NP carriage will be calculated by comparing the proportion of children carrying VT pneumococci 6 months post-vaccination to baseline, at the time of vaccination. The prevalence of colonization of non-VT serotypes will also be described at both timepoints.
Time Frame: During three months of vaccination campaign, and 6 months post-vaccination campaign
Population: Outcome is the percentage of participants with vaccine-type pneumococal carriage in the clusters
Measure: Number; unit: Percentage of participants
Units Other Than Participants: Clusters
Arm/Group | Single Full Dose of PCV 10 | Single Fractional Dose of PCV10 (1/5) | Control Group
Number analyzed (Participants) | 967 | 962 | 321
Number analyzed (Clusters) | 27 | 27 | 9
Percentage of participants | 4.6 | 8.0 | 16.5

2. Secondary Outcome: Vaccine Safety Monitoring
Description: Vaccine safety will be monitored up to 28 days after vaccination and all AEs and SAEs will be recorded.
Time Frame: Up to 28 days after vaccination
Reporting Status: Not Posted

3. Secondary Outcome: Cost-effectiveness and Modeling
Description: An age-structured, dynamic, deterministic model of pneumococcal transmission will be constructed to estimate the impact of mass fractional dose PCV campaigns on VT carriage. The model will use the data on social interactions between age groups and PCV coverage estimates collected during the baseline survey as well as the results of the VT carriage from the baseline survey. Based on the modeled epidemiological impact of PCV10 mass campaigns, with both full and fractional doses, a cost-effectiveness analysis will be performed to estimate the incremental cost-effectiveness ratio of routine PCV10 mass campaigns. The modeled epidemiological impact and cost-effectiveness of a fractional dose mass campaign will be used to inform ongoing discussions of dose-sparing strategies and the use of single-dose fractional PCV in acute humanitarian emergencies.
Time Frame: Within 2 years of study start.
Reporting Status: Not Posted

4. Secondary Outcome: Facilitators and Barriers to Implementing Mass Campaigns of Fractional Dose PCV
Description: A qualitative study will be conducted among parents, healthcare workers, national and international stakeholders to develop insights and recommendations on how a potential future fractional dose PCV mass campaign could be successfully planned, communicated, delivered and integrated into national immunization programs.
Time Frame: Within 2 years of study start.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 28 days following vaccination.
Description: Population under surveillance for adverse events is the total population aged 1-9 living in the 63 clusters.
Arm/Group | Single Full Dose of PCV 10 | Single Fractional Dose of PCV10 (1/5) | Control Group
All-Cause Mortality (participants affected / at risk) | 3/20091 | 4/18821 | 1/5706
Serious Adverse Events (participants affected / at risk) | 28/20091 | 33/18821 | 19/5706
Other Adverse Events (participants affected / at risk) | 0/20091 | 0/18821 | 0/5706
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Full Dose of PCV 10 (N=20091) | Single Fractional Dose of PCV10 (1/5) (N=18821) | Control Group (N=5706)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2) | 5 (5) | 1 (1)
Malaria (Infections and infestations) | 18 (18) | 22 (22) | 13 (13)
Mucocutaneous candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1) | 2 (2)
Respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Kwashiorkor (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 2 (2)
Marasmus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-28): https://cdn.clinicaltrials.gov/large-docs/14/NCT05175014/Prot_SAP_000.pdf